CLINICAL TRIAL: NCT00903227
Title: A Proof Of Concept Study To Assess The Steroid Sparing Effect Of Combined Nasal And Inhaled Corticosteroid In Patients With Asthma And Persistent Rhinitis
Brief Title: Steroid Sparing Effect of Nasal Corticosteroid In Asthma And Rhinitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Dundee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NAI03; 2005-005557-22 (EudraCT Number)
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Last update posted 2019-10-16 (Actual); Status verified 2019-10

CONDITIONS: Asthma; Allergic Rhinitis
Keywords: Asthma; Allergic rhinitis; fluticasone; methacholine
MeSH Terms: conditions — Asthma; Rhinitis, Allergic | interventions — Fluticasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Low Dose (Experimental): One puff of inhaled Fluticasone Evohaler pMDI 50 µg twice a day (Total FP dose 100 µg) and 1 puff of inhaled Placebo twice a day with placebo intranasal spray 2 squirts each nostril once a day.
  Interventions: Drug: Fluticasone Evohaler pMDI; Drug: Placebo; Drug: Placebo intranasal spray
- Combined (Experimental): One puff of inhaled fluticasone propionate Evohaler pMDI 50 µg twice a day (Total daily FP dose 100 µg) and 1 puffs of Placebo twice a day with intranasal fluticasone propionate (Flixonase®) 50ug 2 squirts each nostril once a day (i.e. total intranasal FP daily dose 200ug).
  Interventions: Drug: Fluticasone Evohaler pMDI; Drug: Placebo; Drug: fluticasone propionate (Flixonase®)
- High dose (Experimental): One puff of inhaled Fluticasone Evohaler 250µg twice a day (Total daily FP dose 500µg) and 1 puff of inhaled placebo twice a day with placebo intranasal spray 2 squirts each nostril once a day.
  Interventions: Drug: Placebo; Drug: Fluticasone Evohaler; Drug: Placebo intranasal spray

INTERVENTIONS:
Drug: Fluticasone Evohaler pMDI — One puff of inhaled Fluticasone Evohaler pMDI 50 µg twice a day (Total FP dose 100 µg)
  Arms: Combined; Low Dose
Drug: Placebo — 1 puff of inhaled Placebo twice a day
Drug: Fluticasone Evohaler — One puff of inhaled Fluticasone Evohaler 250µg twice a day (Total daily FP dose 500µg)
  Arms: High dose
Drug: Placebo intranasal spray — placebo intranasal spray 2 squirts each nostril once a day
  Arms: High dose; Low Dose
Drug: fluticasone propionate (Flixonase®) — intranasal fluticasone propionate (Flixonase®) 50ug 2 squirts
  Arms: Combined

SUMMARY:
Up to 40% of patients with asthma have allergic rhinitis and treatment of nasal airway inflammation with topical steroids improves the twitchiness of the airways (hyperresponsiveness) and overall asthma control. The use of inhaled corticosteroids reduces symptoms, severity of asthma attacks, improves quality of life, and reduces asthma related deaths. Similarly, treatment of rhinitis with nasal steroids reduces symptoms and improves quality of life. While there is evidence that combined treatment of the nose and the lungs with topical steroids improves symptoms and underlying inflammation, it is unclear whether such control can be achieved using a smaller dose of inhaled steroid in combination with nasal steroid. It is therefore the intention of this study to evaluate if combination steroid therapy (nose and lungs) has a steroid sparing effect in patients with asthma and rhinitis using sensitive markers of airway inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Mild to moderate atopic asthmatics with FEV1 ≥ 60% on ≤ 1000 ug BDP and concomitant persistent allergic rhinitis (SPT +ve and PC20 < 4 mg/ml)
* Male or female aged 18-65 years
* Informed Consent
* Ability to comply with the requirements of the protocol

Exclusion Criteria:

* Severe asthmatics as defined by an FEV1 ≤ 60% or PEF variability > 30% or with continual daytime or nocturnal symptoms.
* Nasal Polyposis grade 2/3, deviated nasal septum ≥ 50%
* The use of oral corticosteroids within the last 3 months
* Recent respiratory tract infection (2 months)
* Significant concomitant respiratory disease
* Any other significant medical condition or investigation which may jeopardise the safety of the participant or the conduct of the protocol
* Any significant abnormal laboratory result as deemed by the investigators
* Pregnancy, planned pregnancy or lactation
* Known or suspected contra-indication to any of the IMP's
* Concomitant use of medicines (prescribed, over the counter or herbal) that may interfere with the trial

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-12; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
methacholine PC20 | 0, 2, 4, 6, 8, 10, 12 weeks

SECONDARY OUTCOMES:
Spirometry | 0, 2, 4, 6, 8, 10, 12 weeks
Juniper AQLQ | 0, 2, 4, 6, 8, 10, 12 weeks
Fractionated Nitric Oxide | 0, 2, 4, 6, 8, 10, 12 weeks
serum ECP | 0, 2, 4, 6, 8, 10, 12 weeks
blood eosinophils | 0, 2, 4, 6, 8, 10, 12 weeks
Overnight urinary cortisol creatinine | 0, 2, 4, 6, 8, 10, 12 weeks
Peak Nasal Inspiratory Flow rate | 0, 2, 4, 6, 8, 10, 12 weeks
Nasal Nitric Oxide | 0, 2, 4, 6, 8, 10, 12 weeks
Juniper mini RQLQ | 0, 2, 4, 6, 8, 10, 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Arun Nair, MBBS, Principal Investigator — University of Dundee; Brian Lipworth, MD, Study Director — University of Dundee
Locations (1):
- Asthma and Allergy Research Group, Ninewells Hospital and University of Dundee, Dundee, Angus, United Kingdom

REFERENCES:
- [Background] Corren J. Allergic rhinitis and asthma: how important is the link? J Allergy Clin Immunol. 1997 Feb;99(2):S781-6. doi: 10.1016/s0091-6749(97)70127-1. PMID 9042071
- [Background] Reed CE, Marcoux JP, Welsh PW. Effects of topical nasal treatment on asthma symptoms. J Allergy Clin Immunol. 1988 May;81(5 Pt 2):1042-7. doi: 10.1016/0091-6749(88)90177-7. PMID 3131406
- [Background] Dahl R, Nielsen LP, Kips J, Foresi A, Cauwenberge P, Tudoric N, Howarth P, Richards DH, Williams M, Pauwels R; SPIRA Study Group. Intranasal and inhaled fluticasone propionate for pollen-induced rhinitis and asthma. Allergy. 2005 Jul;60(7):875-81. doi: 10.1111/j.1398-9995.2005.00819.x. PMID 15932376
- [Background] Bousquet J, Reid J, van Weel C, Baena Cagnani C, Canonica GW, Demoly P, Denburg J, Fokkens WJ, Grouse L, Mullol K, Ohta K, Schermer T, Valovirta E, Zhong N, Zuberbier T. Allergic rhinitis management pocket reference 2008. Allergy. 2008 Aug;63(8):990-6. doi: 10.1111/j.1398-9995.2008.01642.x. PMID 18691301
- [Result] Nair A, Vaidyanathan S, Clearie K, Williamson P, Meldrum K, Lipworth BJ. Steroid sparing effects of intranasal corticosteroids in asthma and allergic rhinitis. Allergy. 2010 Mar;65(3):359-67. doi: 10.1111/j.1398-9995.2009.02187.x. Epub 2009 Oct 5. PMID 19804441